CLINICAL TRIAL: NCT01786941
Title: Regulation of Branched-chain Amino Acid Metabolism in Pre-Diabetes: Responses to Exercise Training and Gastric Bypass Surgery
Brief Title: Regulation of Branched-chain Amino Acid Metabolism in Pre-Diabetes
Acronym: BCAAM-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00034434
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Branched-chain Amino Acid Metabolism; Insulin Sensitivity
Keywords: Branched-chain Amino Acids; Insulin Sensitivity; Exercise; Leucine
MeSH Terms: conditions — Insulin Resistance; Motor Activity

ARMS (3):
- Lean Group (No Intervention): Healthy Controls - no intervention
- Pre-Diabetes Group (Other): Pre-Diabetes Group will undergo a 6-mo Aerobic and Resistance combined exercise training intervention
  Interventions: Other: Pre-Diabetes Group - 6-mo Aerobic and Resistance combined exercise training
- Gastric Bypass Group (Other): Non-diabetic patients intending to undergo Gastric Bypass surgery
  Interventions: Other: GBP Group - Non-diabetics intending to undergo Gastric Bypass surgery

INTERVENTIONS:
Other: Pre-Diabetes Group - 6-mo Aerobic and Resistance combined exercise training
  Arms: Pre-Diabetes Group
Other: GBP Group - Non-diabetics intending to undergo Gastric Bypass surgery
  Arms: Gastric Bypass Group

SUMMARY:
Elevated circulating levels of certain amino acids (the building blocks of protein) are strongly associated with insulin resistance. This study will investigate the metabolism of these amino acids in individuals with normal glucose metabolism compared to overweight or obese pre-diabetic individuals. The purpose of this study is to determine how elevated levels of the branched-chain amino acids may contribute to the development of insulin resistance and ultimately diabetes. An additional purpose is to determine whether exercise or gastric bypass (GBP) surgery intervention can correct aberrations in branched-chain amino acid metabolism as insulin sensitivity improves. This information will be used to further our understanding of the development of insulin resistance and type 2 diabetes in at-risk populations and potentially improve clinical treatment of such conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age:

  * Lean and Overweight Pre-diabetic (PD) groups: 40-65 years
  * Obese Gastric Bypass (GBP) patients: 30-65 years
* Body Mass Index (BMI) within desired range for group:

  * Lean group: 18.0 - 24.9
  * Overweight PD group: 25.0 - 35.4
  * GBP group: 35.0 - 50.0
* Fasting Plasma Glucose level within desired range for group:

  * Lean: < 99 mg/dL
  * PD: > 105 - < 126 mg/dL
  * GBP: > 99
* Oral Glucose Tolerance Test, 2-hour Plasma Glucose results within desired range:

  * Lean: < 139 mg/dL
  * PD: 140-199 mg/dL
* Low density (LDL) cholesterol: < 190 mg/dL
* Triglycerides: < 600 mg/dL
* Resting blood pressure: <160/90 mmHg
* Inactive: Exercise < two days/week (GBP and PD only);
* Peak oxygen use: > 14.0 - < 40.0 ml/kg/min (PD only)
* Medications: Stable use of all medications for > three months
* Body Weight < 495 lbs

Exclusion Criteria:

* Smoker: Tobacco use within the last 12 months
* Dieting or intending to diet (excluding intention for gastric bypass procedure in GBP group)- Not weight stable for > six months or weight loss exceeding five pounds in last six months
* Use of potential confounding medications, e.g. Niacin containing drugs
* History of diabetes, heart disease or taking medication for those conditions
* History of hypertension (high blood pressure) not controlled with medication
* Pregnant or intending to become pregnant
* Unwillingness to participate in study visits, submit to skeletal muscle biopsies and all other study testing or continuously participate in the exercise training intervention program for six months if in overweight PD group
* Orthopedic limitations, musculoskeletal disease and/or injury
* Allergic to xylocaine
* Inability to give blood continuously through an intravenous catheter
* Unwillingness to exercise at least three times per week at the Duke Center for Living during staff supervised times (PD only)
* Exercise compliance less than 85% in any 6 week period (missing > 3 exercise sessions in a 6 week period)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Changes in Branched-chain Amino Acid Metabolism in Pre-Diabetes at Baseline and post-intervention | Baseline and pre- and post-intervention: 1) Lean Group-Baseline measures only; 2)Pre-Diabetic group - Baseline and 6-months post exercise intervention; 3) GBP group - Baseline and 3-months post Gastric Bypass Surgery
  1. Lean Healthy Controls - Baseline only
  2. Pre-Diabetic Group - Baseline and 6-months post the Aerobic and Resistance combined exercise training intervention
  3. Gastric Bypass Group - Baseline and 3-months post Gastric Bypass surgery

SECONDARY OUTCOMES:
Changes in Insulin Sensitivity at Baseline and post-intervention | Baseline and pre- and post-intervention: 1) Lean Group-Baseline measures only; 2)Pre-Diabetic group - Baseline and 6-months post exercise intervention; 3) GBP group - Baseline and 3-months post Gastric Bypass Surgery
  1. Lean Healthy Controls - Baseline only
  2. Pre-Diabetic Group - Baseline and 6-months post the Aerobic and Resistance combined exercise training intervention
  3. Gastric Bypass Group - Baseline and 3-months post Gastric Bypass surgery

CONTACTS AND LOCATIONS:
Overall Officials: William E. Kraus, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Glynn EL, Piner LW, Huffman KM, Slentz CA, Elliot-Penry L, AbouAssi H, White PJ, Bain JR, Muehlbauer MJ, Ilkayeva OR, Stevens RD, Porter Starr KN, Bales CW, Volpi E, Brosnan MJ, Trimmer JK, Rolph TP, Newgard CB, Kraus WE. Impact of combined resistance and aerobic exercise training on branched-chain amino acid turnover, glycine metabolism and insulin sensitivity in overweight humans. Diabetologia. 2015 Oct;58(10):2324-35. doi: 10.1007/s00125-015-3705-6. Epub 2015 Aug 9. PMID 26254576